CLINICAL TRIAL: NCT02934945
Title: Treatment Efficacy of Budesonide/Formoterol in Cough Variant Asthma and Typical Asthma Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-HXNK-004
Record Dates: First submitted 2016-10-07; First posted 2016-10-17 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-07

CONDITIONS: Bronchial Asthma
Keywords: Budesonide/formoterol; Typical asthma; Cough variant asthma
MeSH Terms: conditions — Asthma; Cough-Variant Asthma | interventions — Budesonide; Formoterol Fumarate; Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- patients with CVA(CVA group) (Other): budesonide 160μg and formoterol 4.5ug,1 inhalation ,twice daily ,for six months
  Interventions: Drug: budesonide 160μg/formoterol 4.5μg
- patients with TA(TA group) (Other): budesonide 160μg and formoterol 4.5ug,1 inhalation ,twice daily ,for six months
  Interventions: Drug: budesonide 160μg/formoterol 4.5μg

INTERVENTIONS:
Drug: budesonide 160μg/formoterol 4.5μg — SMART regimen
  Other Names: Symbicort

SUMMARY:
Bronchial asthma is a common respiratory disease characterized by chronic airway inflammation, which have been affecting about 1-18% of the population in the world, causing tremendous economic burden for the patients and countries. Generally, asthma is a heterogeneous disease, and it could be classified into many types on the basis of symptoms, that is, typical asthma, cough variant asthma, and chest tightness variant asthma etc. Typical asthma (TA) is defined according to the history of repeated respiratory symptoms such as wheeze, shortness of breath, chest tightness, and cough, usually with reversible airflow limitation, airway hyper-responsiveness, and airway remodeling. Cough variant asthma (CVA) is characterized by the single manifestation, recurrent cough, which could be improved after the use of bronchodilators. However, according to different guidelines, it is still controversial on the treatment of CVA and TA. The guidelines of Global Initiative for Asthma(GINA) in 2014 put forward the treatment of TA patients, but did not list the treatment specific to CVA. The guideline of ACCP（American College of Chest Physicians） and cough guidelines of China are proposed to treat the CVA effectively with bronchial diastolic drug. Inhaled corticosteroids (ICS) and leukotriene receptor antagonists are effective for the treatment of CVA. Currently, more and more studies supported that application of ICS combined with bronchial dilation agents is more beneficial to CVA patients. Budesonide/formoterol is a compound of ICS and long-acting beta2-agonist(LABA), which can not only be used as a maintenance medication, but also be used as a relief medication, namely, budesonide/formoterol treatment regimen for SMART (Symbicort as both maintenance and reliever therapy). Most studies show that SMART treatment can be used in the treatment of TA patients. But the study on whether budesonide/formoterol can be used to treat CVA is still little. To provide basis for clinical medication guidance for patients with CVA and TA, this study will enroll 30 patients with TA or CVA , who will be required to adopt the SMART regimen in the following 6 months.The symptom score, airway inflammation, pulmonary function and airway reactivity changes, will be measured every mouth. After the study finished, the investigators will compare the difference between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. aged 15-75
2. first diagnosed corresponding to the diagnostic standards established by Asthma Committee, Respiratory Society, Chinese Medical Association, or previously diagnosed asthma without regular treatment
3. Mch bronchial provocation test is positive
4. the chest X-ray is normal.

Exclusion Criteria:

1. accompanied by other disease of respiratory system
2. combined with serious illness of other system, such as myocardial infarction, severe arrhythmia, malignant tumors and so on
3. women with pregnancy or lactation.

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-01 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Forced Expiratory Volume in first second | up to six months

SECONDARY OUTCOMES:
forced vital capacity | up to six months
Fractional Exhaled Nitric Oxide | up to six months
Asthma Controlled Test | up to six months
Bronchial Provocation Test | up to six months

CONTACTS AND LOCATIONS:
Overall Officials: Huapeng Yu, Ph.D, Study Director — Southern Medical University, China
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China